CLINICAL TRIAL: NCT06991075
Title: A Randomized Controlled Trial of Transcutaneous Electrical Nerve Stimulation for Pain Mitigation During Intrauterine Device Placement
Brief Title: Transcutaneous Electrical Nerve Stimulation for Pain Mitigation During Intrauterine Device Placement
Acronym: TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Michelle Meglin, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00143776
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pain
Keywords: Obstetrics and Gynecology
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TENS (Active Comparator): A TENS 7000 digital TENS unit will be used. A research staff member will apply TENS pads to specified areas on the lower abdomen and lower back corresponding to T10-11 and S2-4 dermatomes. For the active treatment group, the device will be set to 80 Hz (hfTENS) and device intensity (0-8) will be titrated to patient comfort, as is the standard protocol for TENS use.
  Interventions: Device: High frequency transcutaneous electrical nerve stimulation
- Placebo TENS (Placebo Comparator): A TENS 7000 digital TENS unit will be used. A research staff member will apply TENS pads to specified areas on the lower abdomen and lower back corresponding to T10-11 and S2-4 dermatomes. The TENS device will not be turned on.
  Interventions: Device: High frequency transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: High frequency transcutaneous electrical nerve stimulation — TENS 7000 digital TENS unit will be used.

SUMMARY:
Investigators are conducting a study to determine whether high frequency transcutaneous electrical nerve stimulation (hfTENS) is effective at reducing pain in women having an IUD inserted.

DETAILED DESCRIPTION:
The intrauterine device (IUD) is a highly effective contraceptive method with increasing utilization in the last decade. The procedure to both place and remove an IUD is typically performed in the ambulatory gynecologic clinic. Pain associated with IUD insertion is variably described, and evidence suggests that physicians underestimate the severity of pain patients experience with this procedure. Studies have quantified the experience of pain using visual analog scales, demonstrating moderate insertional pain ranging from 5 to 7 out of 10 cm (equivalent to 50-70 out of 100 mm) on VAS. Increasingly, both academic and lay media reports highlight that traumatic nature of a painful IUD placement and call providers to acknowledge and address the pain of IUD placement in a meaningful way.

To date, research has not identified a highly effective strategy to reduce pain during IUD placement. Transcutaneous electrical nerve stimulation (TENS) is a low-cost, low-risk, nonpharmacologic intervention for pain management. The handheld device works by transmitting an electronically generated topical stimulus to a specified area on the body to alter response to pain signals and promote endogenous endorphin release for pain reduction. High frequency TENS (>50 Hz; "hfTENS") significantly reduces pain associated with dysmenorrhea and a range of outpatient gynecologic procedures, including medication abortion, hysteroscopy, and uterine aspiration. This study evaluates an intervention to address pain during IUD placement in the ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form for IUD Insertion
* Stated willingness to comply with all study procedures
* English speaking individuals aged 18 years or older
* Presenting for IUD initiation during ambulatory care visit at MUSC Women's Health
* Opting for either LNG 52mg or copper T380A IUD

Exclusion Criteria:

* Contraindication to IUD initiation (i.e. pregnancy, current pelvic infection, distorted uterine anatomy)
* Contraindication or allergy to ibuprofen
* History of a chronic pain disorder
* Recent opioid use in the previous 30 days
* History of a cardiac arrhythmia
* History of heart disease (i.e. atrial fibrillation, congestive heart failure)
* Presence of an implantable device with an electrical discharge (i.e. pacemaker)
* BMI > 50 (class IV obesity)
* History of TENS use
* Planned pain intervention outside standard of care (i.e. paracervical block, misoprotol) OR preprocedure use of non-standard pain medication (i.e. benzodiazepines, marijuana, muscle relaxers, gabapentin, benadryl)
* History of epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain scores reported at IUD insertion | From enrollment until 5 minutes after procedure completion
  Pain scores at time of IUD insertion as measured by VAS scores between TENS and placebo groups

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC Women's Health- Cannon Street, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will be analyzed according to the statistical plan for manuscript preparation and journal publication. Individual participant data will be shared within the study team including our collaborators at Icahn School of Medicine at Mount Sinai. Also, IPD will be shared with the IRB according to institutional guidelines.